CLINICAL TRIAL: NCT04168957
Title: An Extension Study to Provide Oraxol to Patients Who Completed KX-ORAX-007
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No need to complete the overall survival (OS) follow-up as the sample size was too small to interpret OS.
Sponsor: Athenex, Inc. (Industry)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-008; U1111-1180-5217 (Other: ICTRP)
Record Dates: First submitted 2018-04-13; First posted 2019-11-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Breastcancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oraxol (Experimental): Subjects in KX-ORAX-008 will begin treatment at the last oral paclitaxel dose they received in Study KX-ORAX-007.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — Oraxol (oral paclitaxel + oral HM30181AK-US)
  Paclitaxel: supplied as capsules HM30181 methanesulfonate monohydrate: supplied as HM30181AK-US tablets

SUMMARY:
KX-ORAX-008 is an extension study of patients who completed KX-ORAX-007 without disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and who wish to continue Oraxol treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, extension study offering the option of further Oraxol treatment to breast cancer patients who have completed the KX-ORAX-007 Oraxol study with complete response (CR), partial response (PR), or stable disease (SD), and who wish to continue further Oraxol treatment. The study contains 3 periods: the Screening Period, the Treatment Period, and the Follow-up Period. A Final Visit will occur within 7 days of the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients who have completed Study KX-ORAX-007 without disease progression at Week 16, who wish to continue Oraxol treatment.
2. Signed written informed consent.
3. Willing to fast for 6 hours before and 2 hours after Oraxol administration on all treatment days.
4. Patients must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of assigned study treatment.

Exclusion Criteria:

1. Have not recovered from unacceptable toxicity associated with previous Oraxol treatment in KX-ORAX-007.
2. Are currently receiving other medications intended for the treatment of their malignancy.
3. Women who are pregnant or breastfeeding.
4. Taking any following prohibited medications:

   * Strong inhibitors (eg, ketoconazole) or strong inducers (eg, rifampin or St. John's Wort) of CYP3A4 (within 2 weeks prior to the start of dosing in the study).
   * Strong inhibitors (eg, gemfibrozil) or strong inducers (eg, rifampin) of CYP2C8 (within 2 weeks prior to the start of dosing in the study).
   * Strong P-gp inhibitors or inducers.
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg, digoxin, dabigatran) within 24 hours prior to start of dosing in the study.
5. Use of warfarin. Patients receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements.
7. Known allergic reaction or intolerance to study medication components.
8. Known allergic reaction or intolerance to contrast media.
9. Patients who, in the Investigator's opinion, are not suitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From screening until final visit (within 72 hours prior to Day 21 of Study Period 2, preferably before the participant receives any additional chemotherapy)
  Safety assessments will consist of determining and recording all adverse events and SAEs (adverse events will be graded on a 5-point scale according to CTCAE v4.03); Evaluate the safety of Oraxol. Number of participants with treatment-related adverse events.

SECONDARY OUTCOMES:
Activity: Tumor response | from the start of treatment in KX-ORAX-007 until follow up visit every 2 months after patient withdrawal up to 10 months.
  The number of patients with CR or PR at any post-baseline assessments after the start of treatment in KX-ORAX-007. Computed tomography (CT) and/or magnetic resonance imaging (MRI) scans will be conducted on Day 1 every 8 weeks until documented progression. Tumor status will be evaluated using RECIST v1.1 criteria. In addition to using the RECIST criteria, the Investigator must consider all other clinical information as part of tumor status evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (5):
- Taiwan (5):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Tr-Service General Hospital, Taipei
  - Taipei Veterans Generla Hospital, Taipei, Taiwan, 11217

IPD SHARING:
Plan to Share IPD: Undecided